CLINICAL TRIAL: NCT01446094
Title: Diagnostic Value of a Rapid Protocol Regadenoson Stress Cardiovascular Magnetic Resonance Scan for Detection of Coronary Artery Disease
Brief Title: Diagnostic Study of Rapid Regadenoson Stress Cardiovascular Magnetic Resonance (CMR) to Detect Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dipan Shah (Other)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dipan Shah, Director, Cardiac Magnetic Resonance Imaging, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00006077; IRB(2)0511-0092 (Other: HMRI IRB)
Record Dates: First submitted 2011-09-21; First posted 2011-10-04 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- single-arm (Other): Additional images collected during routine cardiac MRI (CMR) with diagnostic imaging agent, regadenoson.
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — Intravenous administration of 0.4 mg dose of Regadenoson using per routine CMR, as indicated in the package insert.
  Other Names: Lexiscan

SUMMARY:
This study is designed to evaluate the feasibility and diagnostic performance of a novel rapid regadenoson stress CMR protocol for detecting of obstructive coronary artery disease.

DETAILED DESCRIPTION:
This is a single center, open-label, pilot study in subjects scheduled for invasive coronary angiography for evaluation of coronary artery disease. The primary objective is to evaluate the profile of sensitivity, specificity, and diagnostic accuracy of a novel rapid regadenoson stress CMR protocol for detection of >= 70 coronary artery stenosis on invasive coronary angiography. Additionally the objective will be to compare the time for performance of this novel rapid regadenoson stress CMR protocol in comparison to the standard stress CMR protocol.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Scheduled for invasive coronary angiography

Exclusion Criteria:

* Inability to give informed consent
* Possible pregnancy (confirmed by urine test)
* Women who are breastfeeding
* Severe claustrophobia
* Inability to lie flat for 20-30 minutes (the anticipated amount of time to complete the MRI procedure)
* Individuals with cochlear implants
* Individuals with non-MRI compatible aneurysm clips
* Potential contraindications to regadenoson use due to:

Severe lung disease (active wheezing) Severe bradycardia (heart rate < 40 beats/min) Second- or third-degree atrioventricular heart block Sick sinus syndrome History of Long QT syndrome Severe hypotension (systolic BP < 80 mm Hg) Decompensated heart failure

* Contraindication to administration of Gadolinium (Gd) based contrast agents (GBCA):

Stage 4 or 5 chronic kidney disease (eGFR < 30 ml/min/1.73 m2) Known allergy to GBCA

Special Considerations:

- Although individuals who have an occupational history of welding, grinding, or other metal work will not be excluded from the study, they must undergo an orbital x-ray, to exclude any occult metal fragments, before they can participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-08; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Profile of sensitivity, specificity, and diagnostic accuracy of rapid regadenoson stress CMR. | Up to 7 days
  Evaluate the profile of sensitivity, specificity, and diagnostic accuracy of a rapid regadenoson stress CMR protocol for the detection of >= 70% stenosis of a major epicardial coronary artery on invasive coronary angiography.

SECONDARY OUTCOMES:
Evaluate time for performance of rapid regadenoson stress CMR protocol. | Up to 7 days
  Evaluate duration of time for performance of rapid regadenoson stress CMR protocol in comparison to time for performance of standard regadenoson stress CMR protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Dipan Shah, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- The Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan to share data to be determined.

REFERENCES:
- [Background] Wagner A, Mahrholdt H, Holly TA, Elliott MD, Regenfus M, Parker M, Klocke FJ, Bonow RO, Kim RJ, Judd RM. Contrast-enhanced MRI and routine single photon emission computed tomography (SPECT) perfusion imaging for detection of subendocardial myocardial infarcts: an imaging study. Lancet. 2003 Feb 1;361(9355):374-9. doi: 10.1016/S0140-6736(03)12389-6. PMID 12573373
- [Background] Kim HW, Klem I, Shah DJ, Wu E, Meyers SN, Parker MA, Crowley AL, Bonow RO, Judd RM, Kim RJ. Unrecognized non-Q-wave myocardial infarction: prevalence and prognostic significance in patients with suspected coronary disease. PLoS Med. 2009 Apr 21;6(4):e1000057. doi: 10.1371/journal.pmed.1000057. Epub 2009 Apr 21. PMID 19381280
- [Background] Wilke N, Jerosch-Herold M, Wang Y, Huang Y, Christensen BV, Stillman AE, Ugurbil K, McDonald K, Wilson RF. Myocardial perfusion reserve: assessment with multisection, quantitative, first-pass MR imaging. Radiology. 1997 Aug;204(2):373-84. doi: 10.1148/radiology.204.2.9240523.
- [Background] Al-Saadi N, Nagel E, Gross M, Bornstedt A, Schnackenburg B, Klein C, Klimek W, Oswald H, Fleck E. Noninvasive detection of myocardial ischemia from perfusion reserve based on cardiovascular magnetic resonance. Circulation. 2000 Mar 28;101(12):1379-83. doi: 10.1161/01.cir.101.12.1379. PMID 10736280
- [Background] Schwitter J, Nanz D, Kneifel S, Bertschinger K, Buchi M, Knusel PR, Marincek B, Luscher TF, von Schulthess GK. Assessment of myocardial perfusion in coronary artery disease by magnetic resonance: a comparison with positron emission tomography and coronary angiography. Circulation. 2001 May 8;103(18):2230-5. doi: 10.1161/01.cir.103.18.2230. PMID 11342469
- [Background] Nagel E, Klein C, Paetsch I, Hettwer S, Schnackenburg B, Wegscheider K, Fleck E. Magnetic resonance perfusion measurements for the noninvasive detection of coronary artery disease. Circulation. 2003 Jul 29;108(4):432-7. doi: 10.1161/01.CIR.0000080915.35024.A9. Epub 2003 Jul 14. PMID 12860910
- [Background] Klem I, Heitner JF, Shah DJ, Sketch MH Jr, Behar V, Weinsaft J, Cawley P, Parker M, Elliott M, Judd RM, Kim RJ. Improved detection of coronary artery disease by stress perfusion cardiovascular magnetic resonance with the use of delayed enhancement infarction imaging. J Am Coll Cardiol. 2006 Apr 18;47(8):1630-8. doi: 10.1016/j.jacc.2005.10.074. Epub 2006 Mar 27. PMID 16631001
- [Background] Kim RJ, Shah DJ, Judd RM. How we perform delayed enhancement imaging. J Cardiovasc Magn Reson. 2003 Jul;5(3):505-14. doi: 10.1081/jcmr-120022267. PMID 12882082
- [Background] Wu E, Judd RM, Vargas JD, Klocke FJ, Bonow RO, Kim RJ. Visualisation of presence, location, and transmural extent of healed Q-wave and non-Q-wave myocardial infarction. Lancet. 2001 Jan 6;357(9249):21-8. doi: 10.1016/S0140-6736(00)03567-4. PMID 11197356
- [Background] Choudhury L, Mahrholdt H, Wagner A, Choi KM, Elliott MD, Klocke FJ, Bonow RO, Judd RM, Kim RJ. Myocardial scarring in asymptomatic or mildly symptomatic patients with hypertrophic cardiomyopathy. J Am Coll Cardiol. 2002 Dec 18;40(12):2156-64. doi: 10.1016/s0735-1097(02)02602-5. PMID 12505229
- [Background] McCrohon JA, Moon JC, Prasad SK, McKenna WJ, Lorenz CH, Coats AJ, Pennell DJ. Differentiation of heart failure related to dilated cardiomyopathy and coronary artery disease using gadolinium-enhanced cardiovascular magnetic resonance. Circulation. 2003 Jul 8;108(1):54-9. doi: 10.1161/01.CIR.0000078641.19365.4C. Epub 2003 Jun 23. PMID 12821550
- [Background] Gibbons RJ, Abrams J, Chatterjee K, Daley J, Deedwania PC, Douglas JS, Ferguson TB Jr, Fihn SD, Fraker TD Jr, Gardin JM, O'Rourke RA, Pasternak RC, Williams SV; American College of Cardiology; American Heart Association Task Force on practice guidelines (Committee on the Management of Patients With Chronic Stable Angina). ACC/AHA 2002 guideline update for the management of patients with chronic stable angina--summary article: a report of the American College of Cardiology/American Heart Association Task Force on practice guidelines (Committee on the Management of Patients With Chronic Stable Angina). J Am Coll Cardiol. 2003 Jan 1;41(1):159-68. doi: 10.1016/s0735-1097(02)02848-6. No abstract available. PMID 12570960
- [Background] Metz CE, Herman BA, Roe CA. Statistical comparison of two ROC-curve estimates obtained from partially-paired datasets. Med Decis Making. 1998 Jan-Mar;18(1):110-21. doi: 10.1177/0272989X9801800118. PMID 9456215